CLINICAL TRIAL: NCT05969015
Title: Educação em saúde Intensiva na atenção primária à saúde em Pacientes Com Diabetes Mellitus Tipo 2: um Ensaio clínico Randomizado - The Diabetes Care (D-CARE) Study
Brief Title: Intensive Self-care on Glycemic Control in Outpatients With Type 2 Diabetes Mellitus: The Diabetes Care (D-CARE) Study
Acronym: D-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Collaborators: Prefeitura Municipal de Criciúma (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Departamento de Promoção da Saúde (DEPROS), Secretaria de Atenção Primária à Saúde (SAPS) (Unknown); Hospital Universitário São José (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5.011.600
Record Dates: First submitted 2023-07-10; First posted 2023-08-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus
Keywords: Self Management; Behavior; Type 2 Diabetes Mellitus; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus; Behavior

STUDY DESIGN:
Intervention Model Description: This is an effectiveness/pragmatic, parallel-arm, randomized, superiority trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes' assessors will be masked to assigned interventions in all measurements they would perform.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior-changing/Self-Management (Experimental): This arm is composed by group-based interventions aiming to modify the self-management of the patients through the Prochaska and DiClemente transtheorical model. It is composed by weekly meetings, lasting up to 1 hour and a half, targeting eight patients per group. After the 12nd month of intervention, the meetings will be held each fifteen days untill the trial ending (18 months). The meetings will deal with lifestyle matters, such as nutrition, weight management, and physical activity, as well as medication adherence, blood glucose testing, and others. Whenever a care provider will be assigned to a group, he/she will go over untill the final of the trial, unless unexpected motivations appear. Patients achieving maintenance will receive green flag from the group-based interventions to avoid contamination. It is up to the care provider to perceive the readiness of the patient to another stage.
  Interventions: Behavioral: Prochaska and DiClemente transtheorical model
- Usual Care (No Intervention): Patients randomized to the usual care group will follow the same schedule of the experimental group for outcome assessment; however, the trial team will not intervene in the group - i.e., the group will continue their care routine in their primary care unit.

INTERVENTIONS:
Behavioral: Prochaska and DiClemente transtheorical model — The Prochaska and DiClemente model will be combined to a self-management program in patients with T2DM within 18 months. They will be classified accordingly to their readiness for changing. A care provider will manage the group towards an optimal self-management, aiming to improve their glycemic control and other outcomes of relevance. We will conduct 1 session per week until the end of 12nd intervention month. After, the sections will be conducted each 2 weeks until the end of the trial. Healthcare professional will provide support to the care provider. The recommended processes to progress the patients will be used to trigger them accordingly to their stage, at the discretion of the care provider. We will also consider individualities and non-anticipated problems as a part of the process of behavior changing.
  Arms: Behavior-changing/Self-Management

SUMMARY:
Type 2 diabetes mellitus (T2DM) leads to a high burden of morbidity and mortality, usually attributable to cardiovascular (CVD) causes. A major concern about the disease is that the success of the treatment is highly dependent on self-management, which very often incurs the necessity of behavior change. However, modifying such behaviors, usually linked to daily-life activities, is challenging. Then, the investigators aimed to test the optimal self-management that could be achieved in a reasonable manner carried forward through the Prochaska and DiClemente behavior-changing strategy in a follow-up of 18 months, compared to usual care. Our primary outcome is the between-group difference in HbA1c (%) levels.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients diagnosed with type 2 diabetes mellitus - T2DM (HbA1c % - ≥ 6.5%, or taking at least one oral hypoglycaemic agent, or medical diagnosis);
* To be regularly assisted by the Sistema Único de Saúde and to have been saw at least one year before randomization;
* Readiness for behavior-changing within the pre-action stages: pre-contemplation, contemplation and preparation;
* T2DM patient of challenging handling (e.g., frequent hypoglycaemic seizures, cardiovascular disease (CVD), etc.);

Exclusion Criteria:

* Pregnant women;
* People living with HIV/AIDS;
* T2DM patients taking erythropoietin, recent blood loss, recent blood transfusion and severe anaemia;
* T2DM patients with CVD under non-optimized treatment; or those that made any CVD procedure; or CVD event (e.g., myocardial infarction) within three months before randomization;
* T2DM patients with severe eye and retine disease;
* Patients participating in another study simultaneously;
* Patients living with others in the same place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Glycemic control | at 3-monthly intervals during 18 month
  Glycemic control as measured by glycated haemoglobin (HbA1c) levels (%)

SECONDARY OUTCOMES:
Blood Pressure control | at 6-monthly intervals during 18 month
  Blood Pressure control as measured by office systolic and diastolic blood pressure (SBP/DBP in mmHg)
All-cause number of health care settings visits | at 6-monthly intervals during 18 month
  All-cause number of health care settings visits measured by counts
Attributable number of health care settings visits to type 2 diabetes mellitus | at 6-monthly intervals during 18 month
  Attributable number of health care settings visits to type 2 diabetes mellitus measured by counts
Weight | at 6-monthly intervals during 18 month
  Anthropometric variables measured in kg
Height | at 6-monthly intervals during 18 month
  Anthropometric variables -measured in meters
Body mass index | at 6-monthly intervals during 18 month
  Anthropometric variables - kg per square meter
Abdominal circumference | at 6-monthly intervals during 18 month
  Anthropometric variables - measured in centimeters (cm)
Physical activity levels - Guidelines for Data Processing and Analysis of the International Physical Activity Questionnaire (IPAQ) - Short Form | at 6-monthly intervals during 18 month
  There are three levels of physical activity suggested for classifying populations; these are the new proposed levels, which take account of the concept of total physical activity of all domains. The proposed levels are: inactive; minimally active and HEPA activeí health-enhancing physical activity; a highly active category
Depression scores by Hamilton Depression Rating Scale - HDR-S | at 6-monthly intervals during 18 month
  A score of 0-7 is generally accepted to be within the normal range (or in clinical emission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Anxiety scores - Hamilton Anxiety Rating Scale (HAM-A) | at 6-monthly intervals during 18 month
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
MARKERS OF FOOD CONSUMPTION - Food and nutrition surveillance system - Brazil | at 6-monthly intervals during 18 month
  Qualitative assessment of food intake for the previous day.
Number of hypoglycemiants, anti-hypertensives and hypolipidemic drugs | at 6-monthly intervals during 18 month
  Count of hypoglycemiants, anti-hypertensives and hypolipidemic drugs taken by patients
Low density lipoprotein levels - LDL-C | at 3-monthly intervals during 18 month
  Serum LDL-C levels in mg/dL
High density lipoprotein levels - HDL-C | at 3-monthly intervals during 18 month
  Serum HDL-C levels in mg/dL
Total cholesterol levels - TC | at 3-monthly intervals during 18 month
  Serum TC levels in mg/dL
Total triglycerides levels - TG | at 3-monthly intervals during 18 month
  Serum TG levels in mg/dL
Creatinine levels | at 3-monthly intervals during 18 month
  Serum creatinine levels in mg/dL
Diabetes Mellitus knowledge (DKN-A) | at 6-monthly intervals during 18 month
  The measuring scale used is from 0 to 15. A score of one (1) is attributed to the correct answer and of zero (0) for the incorrect answer. A score higher than eight (8) indicates knowledge about diabetes mellitus
Diabetes Attitude Questionnaire (ATT-19) | at 6-monthly intervals during 18 month
  ATT-19 is an instrument that seeks to measure psychological adjustment for diabetes mellitus, developed in response to the need for evaluation of the psychological and emotional aspects of the disease. It contains nineteen items that include six factors: a) DM-associated stress, b) treatment receptivity, c) trust in the treatment, d) personal efficiency, e) health perception, and f) social acceptance, with the answers measured using a five-point Likert scale (completely disagree - score 1; up to completely agree - score 5). The total value of the score can vary from 19 to 95 points. A score higher than 70 indicates a positive attitude toward the disease. In this instrument, attitude is related to the decision of the individual to adopt or not the self-care measures for diabetes control.

OTHER OUTCOMES:
Adverse Events | at 6-monthly intervals during 18 month
  Adverse Events as counts: all-cause mortality, cardiovascular mortality, STEMI and non-STEMI (fatal and non-fatal), heart failure diagnosis, unstable angina hospitalizations, cardiovascular procedures, hospital admission or re-admission, chronic kidney disease, retinopathy diagnosis, falls.

CONTACTS AND LOCATIONS:
Overall Officials: Luciane B Ceretta, PhD, Principal Investigator — Universidade do Extremo Sul Catarinense, The D-CARE Coordinator Committee; Cristiane D Tomasi, PhD, Study Chair — Universidade do Extremo Sul Catarinense, The D-CARE Coordinator/Steering Committee; Vanessa IA Miranda, PhD, Study Director — Universidade do Extremo Sul Catarinense, The D-CARE Coordinator/Steering Committee; Andriele Vieira, PhD, Study Director — The D-CARE Steering Committee; Felipe Dal-Pizzol, MD, PhD, Study Director — Universidade do Extremo Sul Catarinense, The D-CARE Adjudication/Medical Committee
Locations (1):
- Universidade do Extremo Sul Catarinense, Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We will work under individual participant data sharing policy in this study. Third parties interest in should contact the D-CARE Study staff. The IPD Data Sharing Statement is disclosed clearly to patients in our informed consent and also was approved by the responsible IRB. The data will be shared in a deidentified manner, altogether with dictionaries, glossaries, statistical/analytic codes and materials. Authors should provide a proposal that should include the merit, objectives, ethical duties and a data safety plan. For further details please contact the IPD data-sharing committee of the D-CARE Study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After 6 months after the release of the main report of the study up with no constraints in the upper limit.
Access Criteria: Under the auspicious of the IPD and steering committee of the D-CARE Study.